CLINICAL TRIAL: NCT03868332
Title: Predictors of Subclinical Atherosclerotic Cardiovascular Diseases (ASCVD) in Patients With Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ammar ahmed ammar, principal investigator, Assiut University
Other Study IDs: posacvdpwibd
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- inflammatory bowel diease patients
- normal indivuals

SUMMARY:
Heart disease and failure are the major causes of mortality and morbidity worldwide, despite significant advances in medical technologies in the diagnosis and treatment of the disease. Cardiovascular disease may arise for various reasons including the steadily increasing incidence of obesity, type 2 diabetes, genetic, environmental, dietary and lifestyle factors. Besides all these, there is much evidence suggetsing that inflammation is an important player in the pathogenesis of heart disease, as well as atherogenesis and atherosclerosis.

DETAILED DESCRIPTION:
Heart disease and failure are the major causes of mortality and morbidity worldwide, despite significant advances in medical technologies in the diagnosis and treatment of the disease. Cardiovascular disease may arise for various reasons including the steadily increasing incidence of obesity, type 2 diabetes, genetic, environmental, dietary and lifestyle factors. Besides all these, there is much evidence suggetsing that inflammation is an important player in the pathogenesis of heart disease, as well as atherogenesis and atherosclerosis(1,2). Clinically, patients with rheumatologic diseases have been found to suffer from coronary heart disease; thus, regular monitoring for Cardiovascular disease should be included as a routine assessment for patients with rheumatologic diseases (3). A most common systemic inflammatory disease is inflammatory bowel disease , which is a collection of ulcerative colitis and Crohn's disease, a chronic intestinal disease that may arise due to different factors, and is precipitated by environmental and genetic susceptibility (4,5). Ulcerative colitis and Crohn's disease are characterized by chronic intestinal inflammation, with gastrointestinal symptoms including diarrhea, blood and pus in stools, abdominal pain, fever and weight loss. The incidence of inflammatory bowel disease is on the increase in Canada (6), Europe (7) and Asia (8

). In ulcerative colitis, inflammation is mostly limited to mucosal layer of the colon and involves rectum and other parts of colon (9). On the other hand, Crohn's disease shows characteristic transmural inflammation and fibrosis and occurs as patchy lesions throughout the gastrointestinal tract (10).

Although inflammatory bowel disease is associated with venous vascular problems such as deep venous thrombosis (11), the extent of risk for the patients with inflammatory bowel disease to develop Cardiovascular disease, in particular coronary artery disease is not well understood. inflammatory bowel disease patients have a 2 to 3-fold higher risk of venous thromboembolism than the general population (12), and this risk is high during acute disease flare, as active inflammation tilts the balance between pro-coagulants and anticoagulants, which leads to the characteristic hypofibrinolysis seen in inflammatory bowel disease (13)

ELIGIBILITY:
Inclusion Criteria:

Patients who are diagnosed as ulcerative colitis / Crhon s disease however in activity or in remission attending the the outpatient clinics and inpatient of gastroenterology units of Internal medicine department

Exclusion Criteria:

* Previous history of hypertension , diabetes mellitus, Dyslipidemia
* Previous history of cardiovascular or cerebrovascular events
* Autoimmune , Neoplastic diseases
* Thromboembolic diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: population of the study will be classified into two groups, one with inflammatory bowel disease ,other is healthy volunteers.
  both groups will be investigated for early cardiovascular atherosclerotic changes.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-07-20 (Estimated); Primary Completion 2021-03-20 (Estimated); Study Completion 2021-03-20 (Estimated)

PRIMARY OUTCOMES:
atherosclerotic effects in patients with inflammatory bowel disease | two years duration
  hypertension and ischemic heart disease

CONTACTS AND LOCATIONS:
Overall Officials: Hussien Ahmed EL-Amen, MD, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: No